CLINICAL TRIAL: NCT04873310
Title: Behavior Problems Prevention Using the Online Triple P Parenting Program: Pilot Study of Acceptability and Feasibility
Brief Title: Behavior Problems Prevention Using the Online Triple P Parenting Program
Acronym: TriplePChile
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de los Andes, Chile (Other)
Collaborators: Municipalidad de Lo Barnechea, Chile (Unknown)
Responsible Party: Principal Investigator, Jorge Gaete, Associate Professor, Universidad de los Andes, Chile
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MLB-TripleP-2021
Record Dates: First submitted 2021-04-21; First posted 2021-05-05 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Parenting
Keywords: program; parental competence; behavior problems; emotional problems
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: In all the assessments, the principal investigator and research assistants will be blind to the trial arm where the schools/students were allocated
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Triple P online with professional support (Experimental): In the online version with professional support, the psychologist in charge will have the role of monitoring the autonomous work of the participants during the 8 sessions, as well as answering questions and doubts that the participants may have regarding the program and its implementation.
  Interventions: Other: Triple P online with professional support
- Triple P online without professional support (Experimental): In the version without professional support, the role of the psychologist in charge will be to keep the platform updated so that the person who self-administers the intervention does not have technical problems associated with the platform.
  Interventions: Other: Triple P online without professional support
- Control group (No Intervention): Control group without any intervention.

INTERVENTIONS:
Other: Triple P online with professional support — The psychologist in charge will have the role of monitoring the autonomous work of the participants during the 8 sessions. The psychologist in charge will also verify that the participants are able to complete the online modules week by week, that they understand the contents taught in the module and that they are practicing the tasks and exercises assigned in each of the modules; in addition to generating an action plan in case the participants are not adhering week by week to the self-administration of the program. The follow-up and contact with the families will be carried out by phone and through a weekly email-type messaging system, implemented within the same platform on which the program material is found
  Arms: Triple P online with professional support
Other: Triple P online without professional support — The role of the psychologist in charge will be to keep the platform updated so that the person who self-administers the intervention does not have technical problems associated with the platform.
  Arms: Triple P online without professional support

SUMMARY:
The Triple P program is a comprehensive system of parenting and family support of multilevel preventive intervention, developed for families with members up to 16 years of age, whose objective is to improve parenting skills and prevent or modify dysfunctional parenting practices, thus reducing Family risk factors that affect both child abuse, behavioral problems and emotional problems.

DETAILED DESCRIPTION:
Based on the importance that evidence-based parental interventions have acquired and the need from the health field to provide innovative alternatives that facilitate access to this type of services, parental support programs given through the web emerge. There is evidence that supports the idea that parenting programs taught through the web have an influence on reducing disruptive behaviors in children.

Triple P Online (TPOL) is an adaptation of the Positive Parenting Program, Triple P, a program that has been empirically tested. This adaptation is a parental intervention through the web with self-directed modality, which is based on Level 4 of the Triple P parental program and is configured in 8 interactive sessions with online modules. The topics covered are: 1) What is Positive Parenting, 2) Reinforcing the behavior we want, 3) Teaching new skills, 4) Managing negative behaviors, 5) Managing disobedience, 6) Preventing problems through planning, 7) Making fun outings, 8) Raising confident and competent children.

The main results observed in the implementation of the online Triple P program are (Sanders et al, 2012): reduction of problem child behavior, dysfunctional parenting styles, increasing parents' confidence in their parenting role, and reduction of parental anger.

ELIGIBILITY:
Inclusion Criteria:

* Belong to one of the three socio-economic levels according to SIMCE classification (High, Medium and Low).
* Attend to a primary school of the Municipality of Lo Barnechea, Santiago, Chile.
* Previous participation in the instruments validations stages.
* Identification in The Strengths and Difficulties Questionnaire (SDQ) with behavior problems above the 80th percentile.
* Have Internet access.

Exclusion Criteria:

* Attend to a school that is developing or implementing a manualized program for parents associated with the prevention of behavioral problems
* Participating in a similar study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1920 (Estimated)
Dates: Start 2021-04-06 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Acceptability of the program by parents/main caregivers using the Acceptability Scale (AS) | Inmediately Post-intervention
  A questionnaire exploring the acceptability of the program will be answered by parents/main caregivers of students attending Grade 1 to Grade 4, Primary school, who will participate in the intervention. This questionnaire asks about the parents´opinions about the content of the intervention, strategies used, materials, and performance of the health professional helping in the intervention.The latter is only applicable for parents participating in "Group Triple-p online with professional support". The questionnaire also asks about satisfaction and the helpfulness of the program to improve parenting management. For each statement, the answers can go from 1=Strongly disagree to 5=Strongly agree. A high score means higher acceptably and satisfacción with the program. This is a questionnaire created by the research team.
Feasibility of the program using the Feasibility Inventory (FI) | 6 months
  A register will be used to determine the number of schools initially contacted and the number of schools that accepted to participate; number of parents/main caregivers contacted and that consented and assented to participate in the study at baseline and at follow-up; the number of sessions completed by parents in the platform, the number of telephone contacts delivered by the health professionals, the number of meeting over the phone conducted with parents. This Feasibility Inventory (FI) was created by the research team. This registry will not produce a score, rather it will provide indicators to achievements for several areas of the implementation of the program.

SECONDARY OUTCOMES:
Parenting Scale (PS) | One month
  This 30-item questionnaire measures three dysfunctional discipline styles: Laxness (permissive discipline), Over-reactivity (authoritarian discipline, anger, meanness and irritability) and Verbosity (long reprimands or reliance on talking). The scale has good test-retest reliability (r = .83, .82, and .79, respectively) and has been found to discriminate between parents of clinic and nonclinic children; and to correlate with observational measures of dysfunctional discipline. Each item is answered in a scale of 7 points, according to what are the typical behavior parent perform under each scenario. A total score is computed, ranging from 30 to 210. A high score means parents are choosing more effective strategies to deal with different scenarios.
Parenting Task Checklist (PTC) | One month
  This checklist assesses parents' confidence in successfully dealing with 14 difficult child behaviors like whining and temper tantrums (Behavior Self-efficacy), and in dealing with difficult behavior in 14 different settings such as shopping and having visitors (Setting Self-efficacy).
Alabama Parenting Questionnaire (APQ) | One month
  The APQ measures five dimensions of parenting that are relevant to the etiology and treatment of child externalizing problems: (1) positive involvement with children, (2) supervision and monitoring, (3) use of positive discipline techniques, (4) consistency in the use of such discipline and (5) use of corporal punishment. The project will use the dimensions (1), (3), and (4)., and it will not use the dimension of "(2) supervision and monitoring" because it is not relevant for the target population; and "(5) use of corporal punishment" because it is not the focus of the intervention. The parent form will be used. This questionnaire has 22 items. Each statement is answered from 1= Never to 4 = Often. The score ranges from 22 to 44. a High scores means better parenting skills.
The Strengths and Difficulties Questionnaire (SDQ) | 2 months
  The 25-item SDQ measures perceptions of prosocial and difficult behaviors in children aged 3-16 years. It has good test-retest reliability (r = .85) and has been found to discriminate well between low-risk and high-risk samples. Five scale scores are computed: Emotional Symptoms, Conduct Problems, Inattention/Hyperactivity, Peer Problems, and Prosocial Behavior. The first four sub-scales are included into one scleras of "Total Difficulties".
  Each item is answered from 0=Not true to 2=Certainly true. The score of each sub-scale ranges from 0 to 10. In the case of the Total Difficulties scale, Emotional symptoms sub-scale, Conduct Problems sub-scale, Inattention/Hyperactivity sub-scale, and Peer Problems sub-scale, a high score means more symptoms. In the cae of the Prosocial Behavior scale, a high score means stronger prosocial skills.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de los Andes, Santiago, Las Condes, Chile

IPD SHARING:
Plan to Share IPD: Undecided
Investigators plan to deposit the data collected in this study in the "UK Data Service". Data sharing will never compromise participant privacy, neither schools nor students.

REFERENCES:
- [Result] Sanders MR, Baker S, Turner KM. A randomized controlled trial evaluating the efficacy of Triple P Online with parents of children with early-onset conduct problems. Behav Res Ther. 2012 Nov;50(11):675-84. doi: 10.1016/j.brat.2012.07.004. Epub 2012 Aug 18. PMID 22982082
- [Result] Arnold DS, O'Leary SG, Wolff LS, Acker MM. The Parenting Scale: A measure of dysfunctional parenting in discipline situations. Psychological Assessment. 1993; 5(2), 137-144. https://doi.org/10.1037/1040-3590.5.2.137
- [Result] Goodman R, Scott S. Comparing the Strengths and Difficulties Questionnaire and the Child Behavior Checklist: is small beautiful? J Abnorm Child Psychol. 1999 Feb;27(1):17-24. doi: 10.1023/a:1022658222914. PMID 10197403
- [Result] Sanders MR, Woolley ML. The relationship between maternal self-efficacy and parenting practices: implications for parent training. Child Care Health Dev. 2005 Jan;31(1):65-73. doi: 10.1111/j.1365-2214.2005.00487.x. PMID 15658967